CLINICAL TRIAL: NCT00069654
Title: Dietary Nitrate/Nitrite as Sources of Bioactive Nitric Oxide in Patients With Coronary Artery Disease
Brief Title: Dietary Nitrate and Nitrite to Increase Nitric Oxide in Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mark T. Gladwin, M.D./National Heart, Lung, and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 030312; 03-H-0312
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-18

CONDITIONS: Coronary Arteriosclerosis
Keywords: Endothelium; Atherosclerosis; Vasodilation; Ischemia; Exercise; Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Aneurysm; Ischemia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Procedure: Forearm blood flow study
Procedure: Brachial artery reactivity study
Procedure: Treadmill exercise test

SUMMARY:
This study will determine whether dietary nitrates and nitrites can produce nitric oxide in the body and dilate blood vessels in patients with coronary artery disease. Nitric oxide is normally made by endothelial cells that line blood vessels. It plays an important role in maintaining the normal function of arteries by keeping them open and preventing damage from substances such as cholesterol in the blood stream. Coronary artery disease is caused by atherosclerosis (hardening of the arteries or build-up of cholesterol and scar tissue within the walls of the arteries). Once arteries become clogged, the ability of the endothelium to produce nitric oxide diminishes considerably and may speed up the disease process, leading to shortness of breath, chest pain, and an increased risk of heart attack or stroke.

Patients 21 years of age and older with coronary artery disease may be eligible for this study. Participants will have a medical history and physical examination, electrocardiogram (recording of the electrical activity of the heart), echocardiogram (ultrasound test of the heart), treadmill exercise stress test (see below), and will meet with a dietitian. They will be hospitalized at the NIH Clinical Center on two occasions. For 1 week before each admission, they will follow a diet prescribed by an NIH nutritionist. The diet before one admission will be high in nitrates and nitrites, and the diet before the other admission will be low in nitrates and nitrites. Each admission will last 4 days, during which participants will undergo the following tests:

* Forearm blood flow study: Small tubes are placed in the artery and vein at the inside of the elbow of the dominant arm (right- or left-handed) and a small tube is placed in a vein of the other arm. The tubes are used for infusing saline (salt water) and for drawing blood samples. A pressure cuff is placed around the upper part of the dominant arm, and a rubber band device called a strain gauge is also placed around the arm to measure blood flow. When the cuff is inflated, blood flows into the arm, stretching the strain gauge at a rate proportional to the flow. Maximum grip-strength of the dominant arm is measured with a dynamometer. Forearm blood flow is measured and blood samples are drawn at the following times: 20 minutes after the tubes are placed; during a hand-grip exercise; and 4 minutes after the exercise is completed.
* Brachial artery reactivity study: This test measures h...

DETAILED DESCRIPTION:
Nitric oxide (NO) is a soluable gas continuously synthesized by the endothelium that contributes importantly to vasodilator tone of the coronary and systemic circulations by activating guanylyl cyclase in vascular smooth muscle, causing relaxation. Patients with coronary artery disease, however, have deficient synthesis or increased degradation of NO due to endothelial damage or dysfunction. Reduced NO could contribute to symptoms and progression of coronary artery disease through vasoconstriction, platelet activation, inflammatory cell attachment to the arterial wall, and increased growth of cellular elements of the vessel wall. We have recently determined that nitrite, formed by the auto-oxidation of NO, can be converted to bioactive NO, in part through reactions with deoxyheme proteins that exist not only in red blood cells, but also within the vessel wall. An alternative source of bioactive NO may be via the diet, as nitrates reductases present in oral bacteria. Nitrite may then be converted to NO within the acidic environment in the stomach and absorbed into the bloodstream, or absorbed directly and converted to NO in the bloodstream via reaction with deoxyheme proteins. This study is designed to determine the contribution of daily nitrate/nitrite to NO adducts in blood and to vascular dilator tone assessed directly in the forearm and indirectly through treadmill exercise testing. Findings in this study may have important clinical implications not only in coronary artery disease, but also in other conditions associated with regional endothelial dysfunction and reduced endothelial NO bioactivity (e.g., hypertension, diabetes mellitus, hypercholesterolemia, cigarette smoking, estrogen deficiency), and possibly account for the cardiovascular benefit of diets rich in vegetables shown in epidemiological survey studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adults older than 21 years.

Coronary artery disease established by angiography.

No myocardial infarction within 1 month.

Left ventricular ejection fraction greater than 30%.

No congestive heart failure symptoms within 2 months.

Subject provides written, informed consent.

EXCLUSION CRITERIA:

Significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease) as determined by echocardiography.

Subject physically unable to perform treadmill exercise due to neurologic or orthopedic conditions.

Hypersensitivity to organ nitrates.

Insulin-dependant diabetes mellitus.

Coumadin therapy (because of vitamin K content of green leafy vegetables).

Women of childbearing age unless recent pregnancy test is negative.

Lactating women.

Unwillingness to adhere to dietary requirements or allergy to necessary components of diets, as determined during interview by the dietician.

Surgical or disease-related diminished acid secretion.

Significant non-cardiac disease.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2003-09-25; Primary Completion 2009-05-18 (Actual)

PRIMARY OUTCOMES:
Comparison of forearm blood flow during exercise after 3 days of the nitrate-nitrite-enriched diet to forearm blood flow during exercise after 3 days of the nitrate/nitrite-restricted diet. | Measured on day 4 of the nitrite/nitrate enriched and restricted diet

SECONDARY OUTCOMES:
Comparison of effects of high versus low nitrate/nitrite diets on exercise forearm blood flow between the two cohorts of patients. | Measured on day 4 of the nitrite/nitrate enriched and restricted diet.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Palmer RM, Ferrige AG, Moncada S. Nitric oxide release accounts for the biological activity of endothelium-derived relaxing factor. Nature. 1987 Jun 11-17;327(6122):524-6. doi: 10.1038/327524a0. PMID 3495737
- [Background] Palmer RM, Ashton DS, Moncada S. Vascular endothelial cells synthesize nitric oxide from L-arginine. Nature. 1988 Jun 16;333(6174):664-6. doi: 10.1038/333664a0. PMID 3131684